CLINICAL TRIAL: NCT04531475
Title: A Multicenter, Randomized, Double-blind, Double-simulation, Active Comparator-controlled, Parallel-group Phase II Clinical Study to Evaluate the Efficacy and Safety of X842 Capsules at Different Dosages in Patients With Reflux Esophagitis
Brief Title: Study to Evaluate the Safety and Efficacy of X842 in Patients With Reflux Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Sinorda Biomedicine Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SND-X842-201
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Reflux Esophagitis
Keywords: X842; Reflux Esophagitis; GERD; PCAB
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Intervention Model Description: After completing the relevant laboratory tests and endoscopic examinations at screening, subjects who meet the inclusion criteria and do not meet the exclusion criteria are randomly assigned to X842 capsule low-dose group, X842 capsule high-dose group, and lansoprazole enteric-coated capsule group for 4-week treatment and then receive endoscopy. In the study, the duration of subjects receiving treatment with the test drug or comparator is 4 weeks. If a subject has the reflux esophagitis (RE) uncured under endoscopy at week 4 of treatment, the sponsor will give the subject lansoprazole enteric-coated capsules for free for another 4 weeks' treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial uses a double-blind double-dummy design, where both the investigator and the subject are blinded to the drug given to the subject. X842 capsules (test group), lansoprazole enteric-coated capsules (control group), and placebo are provided by the sponsor. The physical appearance, shape, specification and dosage of the test drug and comparator as well as the placebo are generally similar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- X842 50 mg QD (Experimental): X842 50 mg, capsule, orally, once daily and lansoprazole placebo-matching capsule, orally, once daily up to 4 weeks.
  Interventions: Drug: X842; Drug: Lansoprazole Placebo
- X842 100 mg QD (Experimental): X842 100 mg, capsule, orally, once daily and lansoprazole placebo-matching capsule, orally, once daily up to 4 weeks.
  Interventions: Drug: X842; Drug: Lansoprazole Placebo
- Lansoprazole 30 mg QD (Experimental): Lansoprazole 30 mg, capsule, orally, once daily and X842 placebo-matching capsule, orally, once daily up to 4 weeks.
  Interventions: Drug: X842 Placebo; Drug: Lansoprazole

INTERVENTIONS:
Drug: X842 — X842 capsules
  Other Names: Undecided
  Arms: X842 100 mg QD; X842 50 mg QD
Drug: X842 Placebo — X842 placebo-matching capsules
  Other Names: Undecided
  Arms: Lansoprazole 30 mg QD
Drug: Lansoprazole — Lansoprazole capsules
  Other Names: Undecided
  Arms: Lansoprazole 30 mg QD
Drug: Lansoprazole Placebo — Lansoprazole placebo-matching capsules
  Other Names: Undecided
  Arms: X842 100 mg QD; X842 50 mg QD

SUMMARY:
The purpose of the study is to investigate the efficacy and dose-effect relationship of X842 capsules at different dosages in the treatment of reflux esophagitis for 4 weeks in comparison with lansoprazole enteric-coated capsules.

DETAILED DESCRIPTION:
It is designed as a multicenter, randomized, double-blind, double-simulation, high and low dose group, active comparator-controlled, parallel-group study to investigate the efficacy and dose-effect relationship of X842 capsules at different dosages in the treatment of reflux esophagitis for 4 weeks in comparison with lansoprazole enteric-coated capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 years ≤ age ≤ 75 years;
2. Within 14 days prior to randomization, the subjects are endoscopically diagnosed with reflux esophagitis from Los Angeles (LA) grade A to D (notes: the percent of the subjects with LA grade A of RE should be no more than 60% of the all subjects who are planned to be enrolled in the study);
3. Subjects fully understand the trial contents, participate in the trial voluntarily, and sign the informed consent forms.

Exclusion criteria:

1. Subjects who receive X842 capsules or other P-CAB drugs in previous clinical studies;
2. Subjects known to be allergic to X842 capsules or lansoprazole enteric-coated capsules, or relevant excipients of X842 capsules or lansoprazole enteric-coated capsules, such as lactose, microcrystalline cellulose, croscarmellose sodium, sodium dodecyl sulfate, sodium stearyl fumarate, and silicon dioxide;
3. Subjects unable to receive upper gastrointestinal endoscopy;
4. Subjects unable to independently complete the subject diary cards;
5. Subjects known to have any concomitant disease that may affect the esophagus (eosinophilic esophagitis, esophageal varices, dermatosclerosis, viral or fungal infectious esophagitis, or esophageal stenosis), or have a history of esophageal radiotherapy or cryotherapy (but subjects are eligible for this study if they have concomitant esophageal hiatal hernia)
6. Subjects known to have a history of Barrett's esophagus, or who have Barrett's esophagus discovered during endoscopy at screening;
7. Subjects who have acute upper gastrointestinal hemorrhage within 4 weeks prior to enrollment;
8. Subjects with active peptic ulcer discovered during upper gastrointestinal endoscopy, or subjects with suspicious or definite malignancies;
9. Subjects known to have Zollinger-Ellison syndrome or inflammatory bowel disease (IBD);
10. Subjects with concomitant cholecystolithiasis, gallbladder wall crystal or gallbladder polyp discovered by B ultrasonography at screening;
11. Subjects with a history of surgery that may affect the esophagus (for example, fundoplication and mechanical distension for esophageal stenosis), or subjects with a history of cholecystectmy or surgery of stomach or duodenum (except endoscopic excision of benign polyps, and except simple suture surgeries such as for gastric perforation);
12. Subjects with a history of malignancies within 5 years prior to screening (a subject can participate in the study if his /her skin basal cell carcinoma or carcinoma in situ of uterine cervix has been cured);
13. Subjects with concomitant serious diseases of central nervous system, cardiovascular system, respiratory system, liver, kidney, gastrointestinal tract, urinary system, endocrine system, or hematological system, and the investigator thinks these diseases may mix the study results up or affect the safety of the subject;
14. Laboratory test results at screening showing that ALT or AST is larger than 1.5 times of the upper limit of normal, or kidney function index Cr is larger than the upper limit of normal (a re-examination is permitted in the study, and subjects will be excluded if they still fail to meet the inclusion criteria);
15. Subjects who use proton pump inhibitors (PPIs), P-CABs, histamine2 receptor antagonists (H2RAs), or gastric mucosal protectors (except hydrotalcite) within 2 weeks prior to randomization;
16. Subjects who chronically use (>12 doses / month) non-steroidal anti-inflammatory drug (including cyclooxygenase-2 inhibitor), anti-platelet drug (such as aspirin and clopidogrel), or anticoagulant (such as Warfarin) prior to randomization, and can not stop the medication during the trial;
17. At screening, subjects with clinically significant ECG abnormalities, including serious arrhythmia, multifocal preventricular contraction (PVC), grade II or above atrioventricular block, and prolongation of the Q-T interval (QTc≥450 ms in males and QTc≥470 ms in females);
18. Diabetic subjects with poorly controlled blood glucose level (fasting blood glucose (FBG) > 10.0 mmol/L), or hypertensive subjects with poorly controlled blood pressure (systolic pressure ≥150 mmHg or diastolic pressure ≥100 mmHg);
19. Subjects with known acquired immunodeficiency syndrome (AIDS);
20. Subjects who are using atazanavir sulfate or ripivirin hydrochloride at screening;
21. Subjects with a history of long-term abuse of drug or alcohol within 6 months prior to screening;
22. Female subjects with suspicious or known pregnancy, those in breast-feeding period, or those who are planned to become pregnant during the trial. At the investigator's discretion, women of childbearing age who cannot use a medically-proven and reliable method of contraception from signing the informed consent forms to 4 weeks after the last dose of the study;
23. Subject who plan to have a surgery requiring hospitalization, or subject who need to have a surgery during his/her participation in the study;
24. Subjects who participate in other drug/medical device clinical studies and use the drug/medical device within 3 months prior to randomization;
25. Subjects who are considered unsuitable for participating in this trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects Whose Reflux Esophagitis is Cured as Confirmed by Endoscopy at Week 4 of Treatment | 4 weeks
  Subjects cured of RE are defined as subjects who are endoscopically confirmed to be cured of RE.

SECONDARY OUTCOMES:
Proportion of Subjects Whose Reflux Esophagitis LA Grade is Decreased by ≥1 as Confirmed by Endoscopy at Week 4 of Treatment | 4 weeks
  The endoscopic results must describe RE severity according to the LA grading criteria.
Changes in Gerd-Q Score at Week 2 and 4 Compared With the Baseline | Week 2 and Week 4
  Subjects must record RE symptoms that occur within 7d prior to each visit in the Gerd-Q under the guidance of the investigator.
Changes in Serum Gastrin at Week 2 and 4 of Treatment Compared with the Baseline | Week 2 and Week 4
  Serum gastrin testing will be conducted at the central laboratory. The change between the serum gastrin values collected at Weeks 2 and 4 relative to baseline.
Measurement of the PK Profile | Week 2 and Week 4
  Plasma concentrations of X842 and its metabolites are measured to determine X842 exposure in patients.
Number of Subjects Reporting Who Had One or More Treatment-emergent Adverse Event (TEAE) | Up to 6 weeks
  Adverse event is defined as any adverse medical event that is observed in a subject who is receiving a drug treatment or in a clinical study, and that does not necessarily have a causal relationship with the treatment.
Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of blood serum | Up to 6 weeks
  Number of subjects with any markedly abnormal values in laboratory tests of blood serum collected throughout study is reported.
Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of blood | Up to 6 weeks
  Number of subjects with any markedly abnormal values in laboratory tests of blood collected throughout study is reported.
Number of Subjects With Markedly Abnormal Clinical Laboratory assessment of urine | Up to 6 weeks
  Number of subjects with any markedly abnormal values in laboratory tests of urine collected throughout study is reported.collected throughout study is reported.
Number of Subjects With Markedly Abnormal Electrocardiogram (ECG) Findings | Up to 6 weeks
  The investigator or the sub-investigator interpreted the ECG using one of the following categories: "within normal limits", "abnormal but not clinically significant", or "abnormal and clinically significant".
Vital signs of body temperature | Up to 6 weeks
  °C = degrees Celsius
Vital signs of blood pressure | Up to 6 weeks
  Blood pressure measurements included systolic (mmHg) and diastolic (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Pingsheng Hu, Ph.D, Study Chair — Jiangsu Sinorda Biomedicine Co., Ltd
Locations (16):
- China (16):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Liuan People's Hospital, Liu‘an, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Affiliated Hospital of Guzihou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Affiliated Hospital of Xiangnan University, Chenzhou, Hunan
  - The First people's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangxi PingXiang People's Hospital, Pingxiang, Jiangxi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Chongqi Medical University, Chongqing, Sichuan
  - Taizhou Municipal Hospital, Taizhou, Zhejiang
  - Beijing Luhe Hospital Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu S, Han M, Zong Y, Meng F, Liu Q, Tuo B, Zhang Z, Wang Q, Liu X, He S, Zhen Y, Shao D, Wang S, Xu B, Li X, Tang H, Miu Y, Liu C, Hu J, Hu P, Xiu J, Lu M, Wu Y, Zhang S. A Randomized, Comparative Trial of a Potassium-Competitive Acid Blocker (X842) and Lansoprazole for the Treatment of Patients With Erosive Esophagitis. Clin Transl Gastroenterol. 2025 Apr 1;16(4):e00803. doi: 10.14309/ctg.0000000000000803. PMID 39836012